CLINICAL TRIAL: NCT03483545
Title: An Exploratory Study to Evaluate a Mixed Protocol of Menopur (Highly Purified Human Menopausal Gonadotropin) and REKOVELLE (Follitropin Delta) for Controlled Ovarian Stimulation in IVF (in Vitro Fertilization)
Brief Title: Menopur And Rekovelle Combination Study
Acronym: MARCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr François Bissonnette (Industry)
Collaborators: Create Fertility Center (Other); Olive Fertility Centre (Other); Hannam Fertility Centre (Unknown)
Responsible Party: Sponsor-Investigator, Dr François Bissonnette, Principal Investigator, Clinique Ovo
Organization: Clinique Ovo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 000324
Record Dates: First submitted 2018-03-08; First posted 2018-03-30 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Fertility Disorders
Keywords: Ovarian Response; In vitro fertilization; Controlled ovarian stimulation
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follitropin delta and HP-hMG (Experimental): Follitropin delta combined with highly purified human menopausal gonadotrophin
  Interventions: Combination Product: Follitropin delta and HP-hMG

INTERVENTIONS:
Combination Product: Follitropin delta and HP-hMG — Follitropin delta dose will be determined by AMG and weight in Kg. Highly purified human menopausal gonadotrophin will be determined by follitropin delta dose and body weight in Kg

SUMMARY:
This study proposes to evaluate the effect of adding HP-hMG (Menopur) to follitropin delta in a "mixed protocol" regimen, using an individualized, fixed dose of follitropin delta based on the established algorithm, combined with a variable, adjustable dose of Menopur based on body weight and ovarian reserve.

DETAILED DESCRIPTION:
The initial dose of follitropin delta will be determined at enrolment by the analysis of serum AMH on days 2 to 5 of the menstrual cycle preceding the IVF treatment cycle and body weight in Kg The initial dose of HP-hMG to be added on top of follitropin delta will be determined at enrolment by the total follitropin delta dose and body weight in Kg

ELIGIBILITY:
Inclusion Criteria:

* Women 18 to 40 years of age undergoing their first IVF/ICSI cycle
* Diagnosed with unexplained infertility, tubal infertility, endometriosis stage I/II, or with partners diagnosed with male factor infertility
* Regular menstrual cycles of 24-35 days
* Presence of both ovaries
* Early follicular phase FSH serum concentration <10 IU/L measured between Day 2 to Day 5 of menstrual cycle within the previous 12 months
* Ejaculated sperm (fresh or frozen) for insemination

Exclusion Criteria:

* Inability to consent
* Endometriosis stage III and IV
* High risk of OHSS (AMH ≥ 35 pmol/L)
* History of recurrent miscarriages defined as ≥ 3 consecutive losses
* Women undergoing egg donation
* Women participating in any other research project
* Use of hormonal preparations (except for thyroid medication) during the last menstrual cycle
* Hypersensitivity to follitropin delta and/or HP-hMG

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of utilizable blastocysts on Day 5 or Day 6 of embryo culture | 6 days of embryo culture
  Utilizable blastocyst is defined as embryo at day 5 or 6 suitable for transfer

SECONDARY OUTCOMES:
Determine dosage of REKOVELLE and Menopur in a mixed protocol | up to 20 days
  Evaluate the effect of adding HP-hMG (Menopur) to follitropin delta (REKOVELLE) during IVF stimulation
Evaluate the safety profile of the REKOVELLE - Menopur mixed protocol algorithm | up to 20 days
  The safety profile is the proportion of women with early and late OHSS and/or preventive interventions for early OHSS (i.e., triggering with GnRH agonist, use of dopamine agonist, conversion of planned fresh transfer into a freeze-all). OHSS is defined as an iatrogenic complication that occurs mainly due to ovarian overstimulation by gonadotropins.

CONTACTS AND LOCATIONS:
Overall Officials: François Bissonnette, MD, Principal Investigator — Clinique Ovo; Clifford Librach, MD, Principal Investigator — CReATe Fertility Centre; Tom Hannam, MD, Principal Investigator — Hannam Fertility Centre; Al Yuzpe, MD, Principal Investigator — Olive Fertility Centre
Locations (4):
- Canada (4):
  - Olive Fertility Centre, Vancouver, British Columbia
  - Hannam Fertility Centre, Toronto, Ontario
  - CReATe Fertility Centre, Toronto, Ontario
  - Clinique Ovo, Montreal, Quebec

REFERENCES:
- [Derived] Bissonnette F, Minano Masip J, Kadoch IJ, Librach C, Sampalis J, Yuzpe A. Individualized ovarian stimulation for in vitro fertilization: a multicenter, open label, exploratory study with a mixed protocol of follitropin delta and highly purified human menopausal gonadotropin. Fertil Steril. 2021 Apr;115(4):991-1000. doi: 10.1016/j.fertnstert.2020.09.158. Epub 2020 Nov 30. PMID 33267959